CLINICAL TRIAL: NCT00056433
Title: Evaluation of Potential Synergy of Combining Hydroxyurea With Nitric Oxide Donors on Fetal Hemoglobin Synthesis in Patients With Sickle Cell Anemia
Brief Title: Evaluation of Hydroxyurea Plus L-arginine or Sildenafil to Treat Sickle Cell Anemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 030127; 03-CC-0127
Record Dates: First submitted 2003-03-12; First posted 2003-03-13 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2015-12-07

CONDITIONS: Sickle Cell Anemia
Keywords: Fetal Hemoglobin Induction; L-Arginine; Nitric Oxide Therapy; Sickle Cell Disease; Sildenafil (Viagra); Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea; Arginine; Sildenafil Citrate

INTERVENTIONS:
Drug: Hydroxyurea
Drug: L-Arginine
Drug: Sildenafil

SUMMARY:
Patients with sickle cell disease have abnormal hemoglobin (the protein in red blood cells that carries oxygen to the body). This abnormality causes red blood cells to take on a sickle shape, producing disease symptoms. Fetal hemoglobin, a type of hemoglobin present in fetuses and babies, can prevent red cells from sickling. The drug hydroxyurea increases fetal hemoglobin production in patients with sickle cell disease by making a molecule called nitric oxide. The drugs L-arginine and Sildenafil (Viagra) increase the amount or the effect of nitric oxide. This study will evaluate:

* The safety of giving L-arginine or Sildenafil together with hydroxyurea in patients with sickle cell disease;
* The effectiveness of L-arginine plus hydroxyurea or Sildenafil plus hydroxyurea in increasing fetal hemoglobin in patients with sickle cell disease; and
* The effectiveness of L-arginine plus hydroxyurea or Sildenafil and hydroxyurea in lowering blood pressure in the lungs of patients with sickle cell disease. (Pulmonary blood pressure is elevated in about one-third of patients with sickle cell disease, and this condition increases the risk of dying from the disease.)

Patients with hemoglobin S-only, S-beta-thalassemia, or other sickle cell disease genotype may be eligible for this study.

Before starting treatment, patients will have a complete medical history and physical examination. All patients will take hydroxyurea once a day every day by mouth for at least 2 months. They will be admitted to the NIH Clinical Center to take their first dose of hydroxyurea, and will have blood drawn through a catheter (plastic tube placed in a vein) every hour for 6 hours for tests to determine nitric oxide levels. After discharge, they will return to the clinic once every 2 weeks to check for treatment side effects and for blood tests to monitor hemoglobin and fetal hemoglobin levels. After fetal hemoglobin levels have been stable for 2 months, patients will be admitted to the Clinical Center for their first dose of L-arginine (for men) or Sildenafil (for women). Again, blood samples will be collected through a catheter once an hour for 6 hours. If there are no complications, patients will be discharged and will continue taking hydroxyurea once a day and L-arginine or Sildenafil three times a day for at least 3 months until fetal hemoglobin levels have been stable for at least 2 months. Patients will return to the clinic for blood tests every week for 2 weeks and then every 2 weeks to monitor hemoglobin and fetal hemoglobin levels and to check for treatment side effects.

Patients will have eye examinations before and during treatment. Some patients with sickle cell disease develop abnormalities in the blood vessels of the eye. Also, Sildenafil can cause temporary changes in color vision. Rarely, more serious eye problems can occur, such as bleeding from the eye blood vessels or damage to the retina a layer of tissue that lines the back of the eye. Patients will also have an echocardiogram (ultrasound of the heart) before beginning treatment, after hydroxyurea treatment, and after 1 and 3 months of combined treatment with hydroxyurea and L-arginine or Sildenafil to help measure blood pressure in the lungs.

Patients who develop complications from L-arginine or Sildenafil may continue in the study on hydroxyurea alone. Patients whose fetal hemoglobin levels increase with the combination therapy of hydroxyurea and L-arginine or Sildenafil may continue to take them.

DETAILED DESCRIPTION:
Hydroxyurea is a cell-cycle specific agent that blocks DNA synthesis by inhibiting ribonucleotide reductase, the enzyme that converts ribonucleotides to deoxyribonucleotides. Hydroxyurea has been shown to induce the production of fetal hemoglobin (HbF), initially in non-human primates, and now in patients with sickle cell anemia. The majority of patients with sickle cell disease respond to the drug with a more than two-fold increase in HbF levels; in some patients the percent of HbF exceeds 10 or 15 percent. It is estimated that levels of 20 percent are required to substantially reduce the sickling propensity of red cells and to modulate disease severity. We have recently found that hydroxyurea therapy is associated with the intravascular and intraerythrocytic generation of nitric oxide (NO), and that NO accounts for HbF induction via the guanylyl cyclase/cGMP dependent pathways. In fact, NO donors such as S-nitroso-cysteine and NONOates similarly induce HbF expression in human erythropoietin treated human CD 34+ stem cells. Possible synergy between NO donor therapy and classic cytostatic and differentiating medications should be explored. We propose to treat several patients chronically with hydroxyurea to determine hematological changes Iongitudinally. Once a maximal Hb-F raising effect of hydroxyurea has been established, oral L-arginine (the substrate for NO synthase) and sildenafil (Viagra, a phosphodiesterase inhibitor that potentates cGMP dependent signaling) will be added to determine the ability of other agents to enhance HbF synthesis, especially in hydroxyurea non-responders or partial-responders. Additionally, we have found that up to 33% of patients with sickle cell disease also have secondary pulmonary hypertension, measured by echocardiogram. A secondary endpoint of this study will be to evaluate if chronic hydroxyurea therapy and the addition of L-arginine or sildenafil will improve the pulmonary hypertension in this subgroup.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients must have documented hemoglobin S-only, S-beta-thalassemia, or other sickle cell disease genotype. Only patients with hemoglobin S-only will be considered in the primary analysis.
  2. Patients must have relatively well preserved renal and hepatic function (creatinine less than 1.6 mg/dl and normal liver function test less than 5 X normal ALT).
  3. Evidence of severe sickle cell anemia will include one or more of the following: recurrent pain crisis (greater than or equal to 2 ER visits per year), recurrent acute chest syndrome (a lung problem like pneumonia), hospitalizations, leg ulceration, priapism, aseptic necrosis of the hip, and/or pulmonary hypertension.
  4. Patients must be able to provide informed consent.

EXCLUSION CRITERIA:

1. Patients who have hemoglobin S and A (trait) or hemoglobin A-only (non-sickle cell).
2. Patients must not be on a chronic transfusion program, defined as regular transfusions every 2-8 weeks.
3. Patients must not be pregnant or breast feeding.
4. Patients on chronic nitrates, such as nitroglycerin.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-03-10; Primary Completion 2006-12-27 (Actual); Study Completion 2006-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rodgers GP, Dover GJ, Noguchi CT, Schechter AN, Nienhuis AW. Hematologic responses of patients with sickle cell disease to treatment with hydroxyurea. N Engl J Med. 1990 Apr 12;322(15):1037-45. doi: 10.1056/NEJM199004123221504. PMID 1690857
- [Background] Goldberg MA, Brugnara C, Dover GJ, Schapira L, Charache S, Bunn HF. Treatment of sickle cell anemia with hydroxyurea and erythropoietin. N Engl J Med. 1990 Aug 9;323(6):366-72. doi: 10.1056/NEJM199008093230602. PMID 1695325
- [Background] Charache S, Dover GJ, Moore RD, Eckert S, Ballas SK, Koshy M, Milner PF, Orringer EP, Phillips G Jr, Platt OS, et al. Hydroxyurea: effects on hemoglobin F production in patients with sickle cell anemia. Blood. 1992 May 15;79(10):2555-65. PMID 1375104